CLINICAL TRIAL: NCT01985815
Title: Refining the Target for Deep Brain Stimulation (DBS) in Severe, Treatment Refractory Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: s50927
Record Dates: First submitted 2013-10-22; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; Deep Brain Stimulation; Psychosurgery
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VC/VS stimulation ON followed by OFF (Experimental): triple blind, randomised, two periods of three months
  Interventions: Device: VC/VS stimulation
- VC/VS stimulation OFF followed by ON (Experimental): triple blind, randomised, two periods of three months
  Interventions: Device: VC/VS stimulation

INTERVENTIONS:
Device: VC/VS stimulation
  Other Names: Neurostimulator: Kinetra (Medtronic); Electrode: 3387 (Medtronic)

SUMMARY:
In select, therapy resistent patients with Obsessive Compulsive Disorder (OCD) Deep Brain Stimulation (DBS) has been used as a treatment. DBS is a therapy modality in which electrodes are implanted within specific sub-structures of the brain in order to modulate the activity in targeted neural circuits associated with different neurological disorders. The results of this novel approach to psychiatric disorders have been optimistic. This study aims to investigate wether or not the distance to target location has an influence on the outcome.

In order to deliver DBS, leads containing four electrodes are implanted into the brain target in the ventral capsule/ventral striatum (VC/VS). After an optimization period, patients enter a triple blind randomised two fazed crossover design of two periods of three months. In both crossover branches, patients, evaluating psychiatrist and psychologist are blinded for the stimulation conditions. These conditions are stimulation ON (at optimal parameters) and stimulation OFF. Stimulation parameters are constant during the entire period. During the second crossover branch, stimulation conditions are reversed for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD following the diagnostic and statistical manual of mental disorders-fourth edition (DSM-IV) criteria for OCD (300.3).
* Failure of documented trials of pharmacotherapy, following an appropriate treatment algorithm for OCD.
* Failure of documented trial of cognitive and behavioural therapy
* Duration of illness: min. 5 year
* Y-BOCS at least 30/40.
* Age: 20-65 year

Exclusion Criteria:

* DSM-IV diagnosis on axis 2 of severe personality disorder in cluster A or B, especially in the case of heightened risk for acting-out behavior.
* DSM-IV diagnosis on axis 3 of organic brain pathology or significant abnormalities on MRI.
* Present or past history of psychotic symptoms.
* Present substance abuse, or instable remission of substance abuses (i.e. no substance abuse during the last 12 months).
* Any disorder affecting cognitive functioning, other than motor tics and Gilles de la Tourette's Syndrome
* Mental retardation. A minimum threshold of cognitive skills is needed for adequate reporting on questionnaires and evaluation, and for technical handling of the instruments in a later faze.
* The patient must be juridical free.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (Y-BOCS) | up to 12 months

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | up to 12 months
Global assessment of functioning (GAF) | up to 12 months
Hamilton scale for anxiety | up to 12 months
Beck depression inventory | up to 12 months
Inventory of Depressive Symptoms (IDS) | up to 12 months
Patient Global Impression (PGI). | up to 12 months
Symptom Checklist (SCL-90) | up to 12 months
Quality of Life and Satisfaction Questionnaire (Q-Les-Q) | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium